CLINICAL TRIAL: NCT00014651
Title: Vapreotide in Pancreas Surgery: A Double-Blind, Placebo-Controlled, Randomized Study of Vapreotide to Prevent Post-Surgical Complications in Patients Undergoing Elective Pancreatic Resection Grant Application Title: Vapreotide to Prevent Complications of Pancreatic Resection
Brief Title: Vapreotide in Treating Patients Undergoing Elective Pancreatic Resection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Teminated by the DSMB because there are no differences between the control group and the Vapreotide group
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Michael G. Sarr, MD, FACS, Mayo Clinic
Purpose: Supportive Care
Other Study IDs: CDR0000068584; P30CA015083 (NIH); MAYO-IRB-B-234-00; MAYO-FDR001827; NCI-G01-1938
Record Dates: First submitted 2001-04-10; First posted 2004-05-05 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Pancreatic Cancer; Perioperative/Postoperative Complications
Keywords: perioperative/postoperative complications; stage I pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Postoperative Complications | interventions — vapreotide

INTERVENTIONS:
Drug: vapreotide
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs such as vapreotide may prevent complications following pancreatic resection. It is not yet known if vapreotide is more effective than no further therapy in preventing side effects of pancreatic resection.

PURPOSE: This randomized phase III trial is studying vapreotide to see how well it works compared to a placebo in preventing complications in patients undergoing surgery for pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of vapreotide versus placebo in reducing postoperative pancreatic complications in patients undergoing elective pancreatic resection. II. Compare the postoperative complications occurring within 45 days after surgery unrelated to the pancreas, days of hospitalization and survival at 45 days after surgery, number of rehospitalizations, and number of postoperative blood units or packed red blood cells administered in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients undergo surgical resection on day 1 and receive vapreotide subcutaneously twice daily on days 1-7. Arm II: Patients undergo surgical resection and receive a placebo as in arm I. Patients are followed at days 28 and 45.

PROJECTED ACCRUAL: A total of 580 patients (290 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Planned elective pancreatic resection due to presumed pancreatic tumor (either proximal or distal pancreatic lesion) or presumed neoplasm of the ampullary or periampullary region Require peri-anastomotic drain(s) near the pancreaticoenterostomy or near the pancreatic stump closure The following are excluded: Emergency surgery of the pancreas (acute pancreatitis, pancreatic trauma) Known chronic pancreatitis (pancreatic cancer with duct obstructive chronic pancreatitis allowed) Need for total pancreatectomy Need for pancreatic transplantation Need for elective pancreatic-cyst anastomosis Need for pancreatic duct drainage operation without resection (pancreatic stents allowed if performed with partial pancreatic resection) Enucleation of a pancreatic neoplasm

PATIENT CHARACTERISTICS: Age: 18 to 90 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL Renal: Creatinine no greater than 2 times upper limit of normal Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No neoadjuvant or postoperative adjuvant chemotherapy from 2 weeks before to 2 weeks after surgery Endocrine therapy: At least 4 weeks since prior somatostatin or somatostatin analogue No other concurrent somatostatin or somatostatin analogues Radiotherapy: No neoadjuvant or postoperative adjuvant radiotherapy from 2 weeks before to 2 weeks after surgery Surgery: See Disease Characteristics Other: No concurrent pancreatic enzyme inhibitors (e.g., antiproteases) No concurrent immunosuppressive agents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2001-03 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Sarr, MD, FACS, Study Chair — Mayo Clinic
Locations (18):
- United States (18):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Moffett Cancer Center (South), Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Taubman Health Care Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin